CLINICAL TRIAL: NCT04722146
Title: A Multi-arm Phase 1b Study of Teclistamab With Other Anticancer Therapies in Participants With Multiple Myeloma
Brief Title: A Study of Teclistamab With Other Anticancer Therapies in Participants With Multiple Myeloma
Acronym: MajesTEC-2
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108927; 64007957MMY1004 (Other: Janssen Research & Development, LLC); 2020-004404-33 (EudraCT Number); 2023-503440-14-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; pomalidomide; Lenalidomide; Bortezomib; nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Regimen A: Teclistamab + Daratumumab + Pomalidomide (Experimental): Participants will receive teclistamab plus daratumumab plus pomalidomide.
  Interventions: Drug: Teclistamab; Drug: Daratumumab; Drug: Pomalidomide
- Treatment Regimen B: Teclistamab + Daratumumab + Lenalidomide + Bortezomib (21-day Cycles) (Experimental): Participants will receive teclistamab plus daratumumab plus lenalidomide plus bortezomib in 21-day cycles.
  Interventions: Drug: Teclistamab; Drug: Daratumumab; Drug: Lenalidomide; Drug: Bortezomib
- Treatment Regimen C: Teclistamab + Nirogacestat (Experimental): Participants will receive teclistamab plus nirogacestat.
  Interventions: Drug: Teclistamab; Drug: Nirogacestat
- Treatment Regimen D: Teclistamab + Lenalidomide (Experimental): Participants will receive teclistamab plus lenalidomide.
  Interventions: Drug: Teclistamab; Drug: Lenalidomide
- Treatment Regimen E: Teclistamab + Daratumumab + Lenalidomide (Experimental): Participants will receive teclistamab plus daratumumab plus lenalidomide.
  Interventions: Drug: Teclistamab; Drug: Daratumumab; Drug: Lenalidomide
- Treatment Regimen F: Teclistamab + Daratumumab + Lenalidomide + Bortezomib (28-day Cycles) (Experimental): Participants will receive teclistamab plus daratumumab plus lenalidomide plus bortezomib in 28-day cycles.
  Interventions: Drug: Teclistamab; Drug: Daratumumab; Drug: Lenalidomide; Drug: Bortezomib

INTERVENTIONS:
Drug: Teclistamab — Participants will receive teclistamab.
  Other Names: JNJ-64007957
Drug: Daratumumab — Participants will receive daratumumab.
  Arms: Treatment Regimen A: Teclistamab + Daratumumab + Pomalidomide; Treatment Regimen B: Teclistamab + Daratumumab + Lenalidomide + Bortezomib (21-day Cycles); Treatment Regimen E: Teclistamab + Daratumumab + Lenalidomide; Treatment Regimen F: Teclistamab + Daratumumab + Lenalidomide + Bortezomib (28-day Cycles)
Drug: Pomalidomide — Participants will receive pomalidomide.
  Arms: Treatment Regimen A: Teclistamab + Daratumumab + Pomalidomide
Drug: Lenalidomide — Participants will receive lenalidomide.
  Arms: Treatment Regimen B: Teclistamab + Daratumumab + Lenalidomide + Bortezomib (21-day Cycles); Treatment Regimen D: Teclistamab + Lenalidomide; Treatment Regimen E: Teclistamab + Daratumumab + Lenalidomide; Treatment Regimen F: Teclistamab + Daratumumab + Lenalidomide + Bortezomib (28-day Cycles)
Drug: Bortezomib — Participants will receive bortezomib.
  Arms: Treatment Regimen B: Teclistamab + Daratumumab + Lenalidomide + Bortezomib (21-day Cycles); Treatment Regimen F: Teclistamab + Daratumumab + Lenalidomide + Bortezomib (28-day Cycles)
Drug: Nirogacestat — Participants will receive nirogacestat.
  Arms: Treatment Regimen C: Teclistamab + Nirogacestat

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of teclistamab when administered in different combination regimen and to identify the optimal dose(s) of teclistamab combination regimens.

ELIGIBILITY:
Inclusion Criteria:

* Have documented initial diagnosis of multiple myeloma according to international myeloma working group (IMWG) diagnostic criteria
* Meet treatment regimen-specific requirements as follows: Treatment Regimen A (teclistamab [tec]-daratumumab [dara]-pomalidomide [pom]) only: Participant has relapsed or refractory multiple myeloma and has received 1 to 3 prior lines of therapy, including exposure to a proteasome inhibitor (PI) and lenalidomide; Treatment Regimen B (tec-dara-lenalidomide [len]-bortezomib [bor]) only: Participant has newly diagnosed or relapsed/refractory multiple myeloma and is naive to treatment with lenalidomide; Treatment Regimen C (tec-nirogacestat [niro]) only: Participant has relapsed or refractory multiple myeloma and has 1) received 3 or more prior lines of therapy or 2) is double refractory to a PI and an immunomodulatory drug (IMiD) and triple exposed to a PI, an IMiD, and an anti-cluster of differentiation (CD)38 monoclonal antibody (mAb); Treatment Regimen D (tec-len) only: Participant has multiple myeloma and has received greater than or equal to (>=) 2 prior lines of therapy, including exposure to a PI, an IMiD, and an anti-CD38 mAb; Treatment Regimen E (tec-dara-len) only: Participant has newly diagnosed multiple myeloma or if previously treated has received 1 to 3 prior lines of therapy, including exposure to a PI and an IMiD; Treatment Regimen F (tec-dara-len-bor) only: Participant has newly diagnosed multiple myeloma
* Have measurable disease at screening as defined by at least one of the following: serum M-protein level >= 1.0 gram/deciliter (g/dL); or urine M-protein level >= 200 milligrams (mg)/24 hours; or light chain multiple myeloma: serum immunoglobulin (Ig) free light chain (FLC) >= 10 milligram/deciliter (mg/dL) and abnormal serum Ig kappa lambda FLC ratio
* A woman of childbearing potential must have a negative serum (beta human chorionic gonadotropin [hCG]) pregnancy test at screening and a negative urine or serum pregnancy test within 24 hours before the start of study treatment administration and must agree to further serum or urine pregnancy tests during the study
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 6 months after the last dose of study treatment

Exclusion Criteria:

* Prior treatment with any therapy that targets B-cell maturation antigen (BCMA): This exclusion does not apply to Treatment Regimen C
* Live, attenuated vaccine within 30 days before the first dose of study treatment
* Received a cumulative dose of corticosteroids equivalent to >= 140 mg of prednisone within the 14-day period before the start of study treatment administration
* Active central nervous system (CNS) involvement or exhibition of clinical signs of meningeal involvement of multiple myeloma. If either is suspected, brain magnetic resonance imaging (MRI) and lumbar cytology are required
* Known to be seropositive for human immunodeficiency virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2027-10-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Incidence of Adverse Events (AEs) | Up to 2 year and 5 months
  An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Number of Participants with AEs by Severity | Up to 2 year and 5 months
  Number of participants with AEs by severity will be reported.
Number of Participants with Abnormalities in Laboratory Values | Up to 2 year and 5 months
  Number of participants with abnormalities in laboratory values (such as serum chemistry, hematology) will be reported.
Number of Participants with Dose-Limiting Toxicity (DLT) | Up to Cycle 2 Day 21 (each cycle is of 28 days for Treatment Regimen A and 21 days for Treatment Regimen B)
  The Dose Limiting Toxicities (DLTs) are based on drug related adverse events and defined as any of the following events: hematological / non hematological toxicity of Grade 3 or higher.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 year and 5 months
  ORR is defined as the proportion of participants who achieve partial response (PR) or better according to the international myeloma working group (IMWG) 2016 criteria.
Very Good Partial Response (VGPR) or Better Response Rate | Up to 2 year and 5 months
  VGPR or better response rate is defined as the proportion of participants who achieve a VGPR or better response (stringent complete response [sCR]+ complete response [CR]+VGPR) according to the IMWG 2016 criteria.
Complete Response (CR) or Better Response Rate | Up to 2 year and 5 months
  CR or better response rate is defined as the proportion of participants who achieve a CR or better response (sCR+CR) according to the IMWG 2016 criteria.
Stringent Complete Response (sCR) Rate | Up to 2 year and 5 months
  sCR rate is defined as the proportion of participants who achieve an sCR according to the IMWG 2016 criteria.
Duration of Response | Up to 2 year and 5 months
  Duration of response is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of progressive disease (PD), per IMWG criteria.
Time to Response | Up to 2 year and 5 months
  Time to response is defined as the time between date of first dose of study treatment and the first efficacy evaluation at which the participant has met all criteria for PR or better.
Serum Concentrations of Teclistamab | Up to 2 year and 5 months
  Serum concentrations of teclistamab will be reported.
Serum Concentrations of Daratumumab | Up to 2 year and 5 months
  Serum concentrations of daratumumab will be reported.
Serum Concentrations of Nirogacestat | Up to 2 year and 5 months
  Serum concentration of nirogacestat will be reported.
Number of Participants with Presence of Anti-Drug Antibodies to Teclistamab | Up to 2 year and 5 months
  Number of participants with anti-drug antibodies to teclistamab will be reported for all treatment regimens.
Number of Participants with Presence of Anti-Drug Antibodies to Daratumumab | Up to 2 year and 5 months
  Number of participants with anti-drug antibodies to daratumumab will be reported for Treatment Regimen A, B, E and F.
Number of Participants with Presence of Anti-Drug Antibodies to Recombinant Human Hyaluronidase PH20 Enzyme (rHuPH20) | Up to 2 year and 5 months
  Number of participants with anti-drug antibodies to rHuPH20 will be reported for Treatment Regimen A, B, E and F.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (27):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Washington University School Of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - St Vincents Hospital Melbourne, Fitzroy
  - Alfred Health, Melbourne
  - Calvary Mater Newcastle Hospital, Waratah
- Belgium (2):
  - UZA, Edegem
  - UZ Gent, Ghent
- France (5):
  - Centre Leon Berard, Lyon
  - CHU Nantes, Nantes
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Institut Universitaire du cancer de Toulouse-Oncopole, Toulouse
- United Kingdom (3):
  - University College Hospital, London
  - The Christie Nhs Foundation Trust, Manchester
  - The Royal Marsden NHS Trust Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency